CLINICAL TRIAL: NCT03518099
Title: Searching Biomarkers of Acute Intestinal Ischemic Injuries
Acronym: Survibio
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A02211-52
Record Dates: First submitted 2018-04-25; First posted 2018-05-08 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Acute Mesenteric Ischemia
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient (Experimental): Any patient admitted for acute abdomen condition with or without ischemic causes.
  Interventions: Biological: blood sampling
- witness (Experimental)
  Interventions: Biological: blood sampling

INTERVENTIONS:
Biological: blood sampling — Two tubes of 5ml of blood will be collected for Serum collection, 3 tubes of 5 ml of blood taken for plasma collection and 2 tubes of 7 ml of blood taken for DNA collection
  Other Names: urine sampling

SUMMARY:
The aim of the SURVIBIO study is to characterize accurate biomarkers for acute mesenteric ischemia, in particular at early stages.

In the study, the development of biomarkers will be based on the analysis of human biological samples from patients and controls that will be conserved in a biological library. Samples will be analysed in the Laboratory for Vascular Translational Sciences (LVTS, Inserm U1148), in the Department of Biochemistry (Pr Puy, Dr Peoc'h), in Paris V university , in Imperial College of London (Pr Dumas), in Jacques Monod Institute and in Maastricht University Medical Center . The candidate markers will be determined according to an a priori method (form markers already described in the literature) and with no a priori strategy using -omics methods.

DETAILED DESCRIPTION:
Acute intestinal ischemic injury (i3), or intestinal infarction, is an extremely severe condition that affects the intestine, with a mortality rate that is over 80%, and with major anatomical and functional consequences for the surviving patients, mainly because of intestinal resections, which are responsible for chronic intestinal failure, long term parenteral nutrition and an important financial impact on public health.

Even though the incidence of i3 is largely underestimated (mainly because of the lack of knowledge of diagnostic), more than 1000 patients have been surveyed in Paris's hospital through Information Systems Medicalization Program (K550) searching in 2014. Furthermore, i3 represents a digestive emergency for which the only known prognostic factors are the precocity of the diagnostic and treatment.

Investigators have opened in January 2016 the first structure for intestinal vascular emergency (SURVI) within the Groups University Hospitals Paris-Nord Val de Seine. This unique and innovative intensive care structure, which is dedicated to the multidisciplinary treatment of acute mesenteric ischemia, doesn't have any equivalent, and allows the constitution of cohorts with biological and tissular bio-banking.

SURVI provides the patients suffering from intestinal ischemia a "gut and life staving strategy", through a multimodal and multidisciplinary management (M3). M3 is based on a simple algorithm and it brings together experts in intestinal and vascular pathologies that come from different medical disciplines, such as gastroenterology, interventional radiology, vascular surgery, digestive surgery, anaesthesiology and cardiology.

Therefore, the therapeutic strategies aim to limit the complications, to protect the viable intestine, and to remove the necrotic intestine.

Beside the therapeutic strategy that is proposed by SURVI, improvement of the clinical treatment needs to be associated with the finding of new diagnostic tools of intestinal ischemia, that will have to be early, sensitive and specific, as it is the case for troponin in the context of myocardium ischemia.

So far, no biomarker that is sensible and specific enough for the early diagnostic of intestinal ischemia has been found. The CT-scan which is the only diagnostic tool that allow investigators to confirm the diagnostic, in theory, presents a lack of sensibility for the early, not complicated and non-occlusive forms of the disease.

The main prognostic factor of acute intestinal ischemia is the precocity of diagnostic and treatment. Indeed, the mortality rate sharply increases with the occurrence of intestinal necrosis. The problem is that the phases of the disease that precede intestinal necrosis are extremely difficult to diagnose without any biomarker that is sensible and specific enough. Therefore, it is of major importance for the clinician to be provided with one or more biomarker that will help to validate or invalidate the diagnostic of intestinal ischemia, in the context of any acute abdomen condition.

The aim of the SURVIBIO study is therefore to characterize biomarkers for early diagnostic of acute mesenteric ischemia.

In the prospective part of the study, the development of biomarkers will be based on analysis of human biological samples from patients and controls that will be conserved in a biological library and that will be analysed in the Laboratory for Vascular Translational Sciences (LVTS, Inserm U1148) and in the Department of Biochemistry (Pr Puy, Dr Peoc'h). Among the candidate markers, investigators will analyse I-FABP (molecule associated with enterocyte damage at the top of the intestinal villi), D-Lactate (which is specific of intestinal E.coli, and which indicates bacterial translocation, when found in the blood), Citrulline (which is a marker of the functional profile of enterocytes) and ischemia-modified albumin.

In addition to this approach to "candidate" markers based on very brief data from the literature, investigators also wish to develop an unconventional approach, combining a medical approach of proteomics, combining tandem spectrometry with MALDI and establishment of cytokine profile via a multi-complex approach to the emergence of new potential diagnostic biomarkers. The profiles obtained for patients with ischemia are available at profiles obtained on "control" patients, unaffected.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years
* Acute abdominal pain requiring an injected abdominal injected CT scan, at best at non-injected / early arterial / portal time
* Admitted or attended in Beaujon and / or Bichat hospitals
* Patient covered by a social security scheme
* Written consent

Exclusion Criteria:

• lack of abdominal CT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Estimated)
Dates: Start 2018-11-16 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
observation of clinical-bio-scanographic pain related to a splanchnic-mesenteric, occlusive or non-occlusive vascular insufficiency, to abdominal CT angiography, in the absence of another identifiable cause | 2 years

SECONDARY OUTCOMES:
mortality and causes | 2 years
Intestinal resection ratio | 2 years
acute intestinal ischemic injury relapse ratio | 2 years
short gut syndrome features | 2 years
persistency of mesenteric ischemia clinical signs or of ischemic gastric stenosis | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Corcos Olivier, Clichy, France

IPD SHARING:
Plan to Share IPD: Yes